CLINICAL TRIAL: NCT02910713
Title: Multicenter, Randomized, Controlled, Single-Masked, Cross-Over Clinical Trial to Evaluate Dry Eye Symptoms With Application of the Oculeve Intranasal Tear Neurostimulator During Exposure to a Controlled Adverse Environment (CAE®)
Brief Title: Evaluation of Dry Eye Symptoms in CAE With Application of Intranasal Neurostimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OCUN-011
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Intranasal Application (Experimental): Intranasal Tear Neurostimulator applied intranasally device (active), intranasal application for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥ 3 at 2 or more consecutive time points in at least one eye during the CAE exposure.
  Interventions: Device: Intranasal Tear Neurostimulator
- Extranasal Application (Sham Comparator): Intranasal Tear Neurostimulator device applied extranasally (control) for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥ 3 at 2 or more consecutive time points in at least one eye during the CAE exposure.
  Interventions: Device: Intranasal Tear Neurostimulator

INTERVENTIONS:
Device: Intranasal Tear Neurostimulator — The device delivers small electrical currents, activating nerves that stimulate the body's natural tear production system.

SUMMARY:
This study evaluates the safety and effectiveness of the Intranasal Tear Neurostimulator applied intranasally (active) compared with the same device applied extranasally (control) relating to symptoms of dry eye exacerbated by the Controlled Adverse Environment model.

DETAILED DESCRIPTION:
Participants will be randomized to a single application sequence, either sequence "A" (intranasal application followed by control application) or sequence "B" (control application followed by intranasal application) using the device. Upon entering the CAE, participants will complete dry eye questionnaires every five minutes and will administer the device either intranasally or extranasally in randomized sequence when a certain level of ocular discomfort has been reached.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe dry eye disease
* Normal lid/lash anatomy, blinking function and closure as determined by the Investigator
* Literate, able to speak English, and able to complete questionnaires independently

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to risk of clinically significant increased bleeding
* Nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Implanted metallic or electronic device in the head, a cardiac demand pacemaker, or an implanted defibrillator
* Corneal transplant in either or both eyes
* A woman who is pregnant, nursing an infant, or planning a pregnancy at the Screening Visit
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Senchyna, Study Chair — Allergan
Locations (3):
- United States (3):
  - Eye Care Institute, Louisville, Kentucky
  - Total Eye Care, PA, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intranasal and Extranasal data for this crossover study are combined because there is only access to combined arm data for this study. The study was acquired from another organization and limited results data are available.
Groups:
- All Participants: Intranasal Tear Neurostimulator device, intranasal or extranasal (control) application for approximately 3 minutes at Day 0 when the participant experienced an Ocular Discomfort Score (ODS) ≥ 3 at 2 or more consecutive time points in at least one eye during controlled adverse environment (CAE) exposure; followed by Intranasal Tear Neurostimulator device, intranasal or extranasal (control) application for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥ 3 at 2 or more consecutive time points in at least one eye during CAE exposure. Randomization determined the order of intranasal or extranasal application.
Period: Overall Study
Arm/Group | All Participants
Started | 185
Safety Population: Entered CAE | 171
Completed | 143 (Completed=Completed both Intranasal and Extranasal applications.)
Not Completed | 42
Not completed — Protocol Violation | 2
Not completed — Subject Choice | 4
Not completed — Received One Application | 10
Not completed — Received Neither Application | 18
Not completed — Enrollment cap | 7
Not completed — Investigator Discretion | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants. Intranasal and Extranasal data for this crossover study are combined because there is only access to combined arm data for this study. The study was acquired from another organization and limited results data are available.
Groups:
- All Participants: Intranasal Tear Neurostimulator device, intranasal or extranasal (control) application for approximately 3 minutes at Day 0 when the participant experienced an Ocular Discomfort Score (ODS) ≥ 3 at 2 or more consecutive time points in at least one eye during CAE exposure; followed by Intranasal Tear Neurostimulator device, intranasal or extranasal (control) application for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥ 3 at 2 or more consecutive time points in at least one eye during CAE exposure. Randomization determined the order of intranasal or extranasal application.
Arm/Group | All Participants
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Application to Post-Application in Eye Dryness Score (EDS) Using a Visual Analog Scale (VAS)
Description: The participant rated their eye dryness (both eyes simultaneously) at all visits and every 5 minutes during CAE exposure by placing a vertical mark on the 100 mm horizontal line to indicate the level of eye dryness. 0 corresponds to "no dryness" and 100 corresponds to "maximal dryness". A negative change from Baseline indicates improvement. A cross-over linear model was used with symptom relief as the response variable; sequence, application location, period, and the application location by period interaction as fixed effects; and participant (sequence) as a random effect.
Time Frame: Pre-application to Post-application on Day 0
Population: Participants from the Full Analysis Set (FAS) Population, all randomized participants who initiated a study application, who received both intranasal and extranasal applications.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 143 | 143
score on a scale | -16.48 (1.692) | -3.12 (1.692)
Statistical Analysis 1: Comparison: Intranasal Application vs Extranasal Application; Test type: Superiority; p < 0.0001, ANOVA — One-sided p-value for the difference between Intranasal and Extranasal; Least Squares Mean Difference = -13.36, 95% CI 2-sided [-17.31 to -9.40], Standard Error of Mean 1.999

2. Secondary Outcome: Change From Pre-Application to Post-Application in the Ora Calibra Ocular Discomfort Scale (ODS) Score
Description: The participant graded their eye discomfort prior to CAE entry, during CAE exposure to threshold, then starting 1 minute after treatment application every 5 minutes in each eye separately using the Ora Calibra ODS where: 0=no discomfort to 4=constant discomfort. Data from the analysis eye was used to determine effectiveness. The analysis eye was defined as the eye that reached the threshold triggering the first application or if both eyes reach the threshold at the same time, the eye with the higher discomfort score or if both eyes are the same, the right eye was used. A negative change from Baseline indicates improvement. A cross-over linear model was used with symptom relief as the response variable; sequence, application location, period, and the application location by period interaction as fixed effects; and participant (sequence) as a random effect.
Time Frame: Pre-application to Post-application on Day 0
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 143 | 143
score on a scale | -0.93 (0.080) | -0.34 (0.080)
Statistical Analysis 1: Comparison: Intranasal Application; Test type: Superiority; p < 0.0001, ANOVA — One-sided p-value for the difference between Intranasal and Extranasal; Least Squares Mean Difference = -0.60, 95% CI 2-sided [-0.80 to -0.40], Standard Error of Mean 0.101

ADVERSE EVENTS:
Time Frame: Day 0
Description: Safety population included all randomized participants who entered the CAE. Intranasal and Extranasal Adverse Event (AEs) data for this crossover study are combined because there is only access to combined arm data for this study. The study was acquired from another organization and limited results data are available.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/171
Serious Adverse Events (participants affected / at risk) | 0/171
Other Adverse Events (participants affected / at risk) | 0/171

LIMITATIONS AND CAVEATS:
Intranasal and Extranasal data for this crossover study are combined because there is only access to combined arm data for this study. The study was acquired from another organization and limited results data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.